CLINICAL TRIAL: NCT03259581
Title: Safety of Transarterial Chemoembolization in Patients With Elevated Bilirubin
Brief Title: Safety of Transarterial Chemoembolization (TACE) in the Setting of an Elevated Bilirubin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS137
Record Dates: First submitted 2017-08-01; First posted 2017-08-23 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma; Bilirubinemia
Keywords: transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hyperbilirubinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transarterial chemoembolization (Experimental): Transarterial chemoembolization
  Interventions: Combination Product: Transarterial chemoembolization

INTERVENTIONS:
Combination Product: Transarterial chemoembolization — Delivery of lipiodol, chemotherapy (Deoxyrubicin), and particles (embosphere particles) to the arteries feeding hepatocellular carcinoma. While both chemotherapy and particles are delivered this is a single procedure in which the chemotherapy is delivered followed immediately by particles.

SUMMARY:
The aim of this study is to evaluate the safety of selective transarterial chemoembolization (TACE) of hepatocellular carcinoma (HCC) in the setting of an elevated total bilirubin, but relatively normal direct bilirubin.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma (HCC)
* Direct or conjugated bilirubin < 3 mg/dl
* Total bilirubin > 3 mg/dl
* Willing and able to provide informed consent
* >18 years of age

Exclusion Criteria:

* Currently pregnant
* Patients who are surgical or ablation candidates as determined by multidisciplinary hepatobiliary tumor conference.
* Arterial anatomy which would preclude selective transarterial chemoembolization
* Patients who have a INR or platelet count which are not correctable to <1.8 and >35,000 respectively
* Patients with extrahepatic metastases
* Patients with portal vein invasion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Procedure related adverse events | 1 month
  Percentage of adverse events following TACE

SECONDARY OUTCOMES:
Radiologic Response | 1 month
  mRECIST response after TACE
Progression free survival | 1, 3, 6, 12, 18, and 24 months
  Liver PFS and overall PFS
Overall survival | 24 months
  Overall survival
Change in Model for end stage liver disease (MELD) | 7 and 30 days
  Change in MELD (MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43) score at 7 and 30 days post TACE
Change in Child Pugh score | 7 and 30 days
  Change in Child Pugh score at 7 and 30 days post TACE

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States